CLINICAL TRIAL: NCT03976219
Title: Measuring Evoked Potentials From the Spinal Cord and Dorsal Root Ganglion
Acronym: ECAPS SCS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Budgetary Issues
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00100055
Record Dates: First submitted 2019-06-04; First posted 2019-06-05 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evoked potentials of ECAPs and SSEPs (Experimental): Patients implanted with a spinal cord stimulator. In this arm, we are measuring the evoked potentials of electric compound action potentials (ECAPs) and somatosensory evoked potentials (SSEPs).
  Interventions: Other: ECAPS Closed Loop SCS

INTERVENTIONS:
Other: ECAPS Closed Loop SCS — The purpose of this study is to determine the feasibility of recording evoked compound action potentials (ECAPs) and somatosensory evoked potentials (SSEPs) from the spinal cord (SC) and Dorsal root ganglions (DRG), and their suitability as feedback signals.

SUMMARY:
The purpose of this study is to determine the feasibility of recording evoked compound action potentials (ECAPs) and somatosensory evoked potentials (SSEPs) from the spinal cord (SC) and Dorsal root ganglions (DRG), and their suitability as feedback signals.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age.
* Subject is able and willing to comply with the schedule and protocol.

For implantation of DRG stimulator;

* Subject has been diagnosed with complex regional pain syndrome (CRPS I or II).
* Subject has had chronic, intractable pain of the groin or lower limbs for at least 6 months.
* Subject is indicated for implantation of an Abbott DRG stimulation system.
* Subject will be undergoing trial implantation of an Abbott DRG stimulation system.

For implantation of SCS;

* Subject has been diagnosed with chronic, intractable pain of the trunk and/or limbs.
* Subject is indicated for implantation of a SCS system.
* Subject will be undergoing implantation of an Abbott lead.
* Subject has had stable neurologic function in the past 30 days.
* Subject is able to provide informed consent.

Exclusion Criteria:

* Subject will be implanted with 3 or more DRG leads.
* Subject is currently participating in a clinical investigation that includes an active treatment arm.
* Subject has exhibited escalating or changing pain condition within the past 30 days as evidenced by physician examination.
* Subject currently has an active implantable device including an ICD, pacemaker, spinal cord stimulator, or intrathecal drug pump.
* Subject is a prisoner.
* Female subject is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Pain level as measured by pain scale | Visit 1, up to 2 hours
  Measured on a scale 0 to 10, with 0 being no pain and 10 being pain as bad as you can imagine.
Evoked response amplitude for ECAPS | Visit 1, up to 2 hours
  Evoked responses averaged across trials for ECAPS, measured in micro Volts
Evoked response amplitude for SSEPs | Visit 1, up to 2 hours
  Evoked responses averaged across trials for SSEPs, measured in micro Volts

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Viventi, PhD, Principal Investigator — Duke University; Nandan Lad, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No